CLINICAL TRIAL: NCT04019171
Title: Interval Exercise Training for Reducing Anxiety in First-Time Inmates
Brief Title: EXercise Training for Reducing Anxiety in First-Time Inmates
Acronym: EXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Principal Investigator, Fabien Legrand, Professor, Université de Reims Champagne-Ardenne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Legrand_19_02
Record Dates: First submitted 2019-07-05; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interval exercise training (Experimental)
  Interventions: Behavioral: exercise training
- waiting list (No Intervention)

INTERVENTIONS:
Behavioral: exercise training — 6 weeks of physical exercise training. 3 sessions per week. Session duration : 40 minutes. Self-regulated exercise intensity using Borg's ratings of perceived exertion (RPE)
  Arms: interval exercise training

SUMMARY:
Clinical trial with 2 arms ("interval exercise training" or "waiting list") aiming at evaluating the anxiolytic effects of a 6 weeks-long exercise training program in first-time prisoners with elevated anxiety symtpoms

ELIGIBILITY:
Inclusion Criteria:

* First-time prisoners ; elevated state anxiety (> 40 on the state anxiety inventory)

Exclusion Criteria:

* Symptoms of and/or known cardiovascular, metabolic, psychiatric, neurological or neurodevelopmental disease

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
change in state anxiety | before and after the 6 weeks of intervention
  pre- to post-intervention change in the State Anxiety Inventory score (STAI; Spielberger et al., 1993). The STAI has 20 items assessed on a 4-point Likert scale ranging from 1 (not at all) to 4 (most intensive). Consequently, the range of possible scores is 20-80.

IPD SHARING:
Plan to Share IPD: No
statistical data (anxiety means and standard deviations before and after intervention) will be available in the form of a scientific paper in an academic journal for the participants in the active group (exercise) as well as for participants in the no intervention group (waiting list). No individual data will be published.

REFERENCES:
- [Derived] Legrand FD, Ory E, Herring MP. Evaluation of a brief interval exercise training (IET) intervention for first-time prisoners with elevated anxiety symptoms. Anxiety Stress Coping. 2020 Sep;33(5):581-589. doi: 10.1080/10615806.2020.1768244. Epub 2020 May 21. PMID 32436724